CLINICAL TRIAL: NCT01088308
Title: Hemodynamic Differentiation of Tachycardia Episodes Using Tissue Perfusion
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No enrollements for more than 6 months in Phase II
Sponsor: Medtronic BRC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TPS1010
Record Dates: First submitted 2010-03-11; First posted 2010-03-17 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Arrhythmias, Cardiac
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm (Experimental): All Patients underwent Intervention.
  Interventions: Procedure: High rate atrial and vetricular stimulation; Procedure: Ventricular Tachycardia induction

INTERVENTIONS:
Procedure: High rate atrial and vetricular stimulation — The right atria and ventricle of the subject will be electrically stimulated at high rate mimicking tachycardia episodes using electrodes placed in the right atria and ventricle.
  Other Names: High rate pacing
Procedure: Ventricular Tachycardia induction — A programmed electrical stimulation protocol will be performed using an electrode placed in the right ventricle.
  Other Names: VT induction

SUMMARY:
This research study is a prospective, single-center, feasibility study designed to assess the possibility to detect hemodynamic changes during tachycardia episodes using tissue perfusion.

DETAILED DESCRIPTION:
This study is being conducted to evaluate the feasibility to detect hemodynamic changes induced by supra-ventricular or ventricular tachycardia (SVT or VT) using tissue perfusion. Patients with a standard indication for either an electrophysiological study or an implantable cardioverter defibrillators(ICD) implant can be included into this study. Tissue perfusion and arterial blood pressure will be monitored and recorded throughout the electrophysiological procedure or ICD implant testing.

The study will be conducted in two consecutive phases. After completion of study phase I the study phase II will commence. Study phase I will be an acute non-invasive study in patients with an indication for an electrophysiological study, in whom tissue perfusion will be measured non-invasively with an epi-cutaneous tissue perfusion sensor. Phase II will be an acute invasive study in patients with an indication for the implantation of an ICD, in whom the tissue perfusion sensor will be placed in the surgically prepared device pocket on the muscular pectoralis or between the muscular pectoralis major and muscular pectoralis minor.

ELIGIBILITY:
Inclusion Criteria:

* Indication for: an electrophysiological study with ventricular stimulation OR the implantation of an implantable cardioverter defibrillator (ICD)
* Patient is at least 18 years old.
* Patient is able and willing to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2010-03; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Change in hemodynamic state during all tachycardia | <3 hours
  The primary objective is to demonstrate for all tachycardia (supra-ventricular and ventricular tachycardia) a 90 % [two sided confidence interval of 75-100 %] agreement between the true hemodynamic state (stable or unstable) derived from arterial blood pressure measurement and the hemodynamic state determined by tissue perfusion

SECONDARY OUTCOMES:
Change in hemodynamic state during SVT | <3 hours
  The secondary objective is to demonstrate for supra-ventricular tachycardia a 90 % [two sided confidence interval of 75-100 %] agreement between the true hemodynamic state (stable or unstable) derived from arterial blood pressure measurement and the hemodynamic state determined by tissue perfusion.

CONTACTS AND LOCATIONS:
Overall Officials: Emilia Stegemann, Dr. med, Principal Investigator — Universitätsklinikum Aachen
Locations (1):
- Universitätsklinikum, Aachen, Germany

IPD SHARING:
Plan to Share IPD: Undecided